CLINICAL TRIAL: NCT01065142
Title: Does Therapeutic Education Improve Heart Failure Patient Quality of Life?
Brief Title: ETIC (Therapeutic Education in Heart Failure)
Acronym: ETIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: GRSP : Groupement Régional de Santé Publique (Unknown); URML : Union Régionale des Médecins Libéraux (Unknown); Ministry of Health, France (Other Government); URCAM : Union Régionale des Caisses d'Assurances Maladies (Unknown); Sanofi (Industry); Groupe Pasteur Mutualité (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CHU-0067; 2009-A01142-55 (Other: Afssaps)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Heart Failure; Quality of Life
Keywords: Heart Failure; Patient Education as Topic; Primary Health Care; Quality of Life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: Therapeutic education — Improve therapeutic education efficiency on life quality of heart failure patients in general practice

SUMMARY:
Use lay language. Background: Heart failure is an increasingly frequent current pathology due to the population aging and the improvement of acute and chronic heart failure management. Heart failure patients have a poor quality of life because of their symptoms (asthenia, dyspnea…) and frequent hospitalizations. Heart failure is an expensive disease: 1.5 % of the health expenses, 85 % in hospital cost with 200 000 hospitalizations in France per year. Previous studies were multidisciplinary interventions and not realistic in a daily practice for a general practitioner. The aim of this project is to integrate therapeutic education for heart failure patients in a current practice. The patient becomes competent to manage his disease and to identify acute heart failure signs.

Main objective: Improve therapeutic education efficiency on life quality of heart failure patients in general practice.

Second objectives: Describe heart failure patient's hospitalizations.

Methods: Cluster randomized controlled clinical trial comparing intervention and control groups with a follow through for 19 months for each patient. A therapeutic education program will be proposed to the heart failure patients in primary care. The intervention group GP will follow a workshop concerning the therapeutic education concepts and the intervention.

Endpoints: Life quality evaluation (SF-36 and Minnesota scales) and number of hospitalizations of patients in each group.

Population: Heart failure patients in stages I, II, and III of NYHA in primary care. Cluster randomized surgeries in Auvergne (France).

Expected results: The therapeutic education allows the patients to improve their quality of life, to be able to detect their illness signs worsening in a early manner, and to contact their doctor if needed. This would limit the acute heart failure due to treatment adaptation or life habits.

DETAILED DESCRIPTION:
General organisation of the study

* Recruitment of the GP: 3 months (from January to March 2010)
* Training of the intervention group GP during a two days workshop in April 2010 on the therapeutic education and the intervention by an expert team
* Patient Inclusions of by GP: 10 months (from April 2010 to January 2011). The included patients will be followed for 19 months. Some patients will be potentially recruited during the 10th month of inclusion, the follow-up period being of 29 months.
* First consultation used to the inclusion:

  * Information to the patient and collection of the patient written agreement (without informing the intervention objectives in the control group).
  * Evaluation of the life quality in both groups with the SF-36 scale (general) and the Minnesota scale (HF specific) written by the patient or his/her main caregiver (wife or husband, a friend...) in the waiting room after the consultation thanks to a closed envelope given by the GP containing the questionnaire and a pre-paid envelope.
* Intervention of the general practitioner to the patients in the scope of a therapeutic education program:

  * In the intervention group: first session (M1) dedicated to the educative diagnosis after one month. Then 4 sessions of standardized therapeutic education and adapted to the patient each three months for one year. One session in M19 will be dedicated to the synthesis of what the patient learnt from these interventions.
  * In the control group: the patient is followed in consultation in the same deadlines without any particular intervention in M1, M4, M7, M10, M13, M19.
* Life quality evaluation of both groups at 0, 7, 13, and 19 months from the beginning of the inclusion filled in by the patient or his/her main caregiver (husband or wife, a friend...) thanks to a closed envelope given by the GP (at the end of his consultation) containing the questionnaire and pre-paid envelope. These documents are filled in the waiting room after the first consultation and at home in the 7 days following the other consultations. The life quality will be evaluated at the inclusion time (M0), during the intervention (M7 and M13) and at distance (M19) from the end of the intervention. The Minnesota score (22, 23) has been chosen because it is validated and specific of life quality of HF patients. The SF-36 score has also been retained as it permits a generic and global evaluation of life quality and because its reliability, validity and responsiveness have been established (24) (25) (26). SF-36 is the most widely evaluated quality of life measure between 1990 and 1999 (27).
* Collection of the number and the duration of hospital readmission for worsening heart failure and for all cause hospital readmission and of the total number of days of hospitalisation during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Investigators: volunteer randomized general practitioners from the Auvergne region in France.
* The GPs will be randomized in cluster, each GP should recruit at least five patients. If several doctors are part of the same surgery, they will be randomized in the same group (intervention or control). The randomization of the GPs will be stratified by department. The GP commit themselves not to talk of the study between them. Each GP knows in which group of the study he belongs as the intervention group comprises a training seminar but the objectives of the study will not be known by the GPs of the control group.
* All the general practitioners in Auvergne (except homeopaths, acupunctures...) will be contacted by mail to inform them about the study and to invite them to participate to it. The volunteer GPs will have to return their written agreement via a pre-stamped envelope to the investigator center with their coordinates. They will be randomized in both groups (intervention and control). After the formation, each GP of the intervention group would have to recruit at least five patients seen in consultation, who could be included and who have given their written agreement. Each week of the inclusion period, the GP will recruit the first patient having the eligibility criteria until the inclusion of at least five patients. The anonymity of the patients will be guaranteed in the participation contract. The data will be anonymized by the investigator GP and will be submitted to the French electronic data liberty commission (Commission Nationale Informatique et Libertés (CNIL)). The patients could quit the study at any time.

Patients: Systolic or diastolic HF patients to the stages I, II and III of the NYHA followed in primary care. These patients will be recruited by the randomized GP in the intervention and control groups. Patients should be over 50 years old (this age limit expelled only few patients with particular pathology).

Exclusion Criteria:

* • Are not included the stage IV, with short life expectancy, with low efficiency hope of the tested measure, who are very few. The systolic and diastolic HF patients are not distinguished because the possible efficiency of the intervention is not HF type dependent a priori.

  * Dementia as Alzheimer disease diagnosed by GP.
  * Already included in another study
  * Incapacity to follow the education sessions (language problem...)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Life quality evaluation of both groups (control and intervention) at 0, 7, 13, and 19 months from the beginning of the inclusion filled in by the patient or his/her main caregiver (husband or wife, a friend...) thanks to a closed envelope given by the GP | at 0, 7, 13 and 19 months from the beginning of the incusion

SECONDARY OUTCOMES:
Collection of the number and the duration of hospital readmission for worsening heart failure and for all cause hospital readmission and of the total number of days of hospitalisation during the follow-up period. | during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Vaillant-Roussel, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Vaillant-Roussel H, Laporte C, Pereira B, De Rosa M, Eschalier B, Vorilhon C, Eschalier R, Clement G, Pouchain D, Chenot JF, Dubray C, Vorilhon P. Impact of patient education on chronic heart failure in primary care (ETIC): a cluster randomised trial. BMC Fam Pract. 2016 Jul 19;17:80. doi: 10.1186/s12875-016-0473-4. PMID 27436289
- [Derived] Vaillant-Roussel H, Laporte C, Pereira B, Tanguy G, Cassagnes J, Ruivard M, Clement G, Le Reste JY, Lebeau JP, Chenot JF, Pouchain D, Dubray C, Vorilhon P. Patient education in chronic heart failure in primary care (ETIC) and its impact on patient quality of life: design of a cluster randomised trial. BMC Fam Pract. 2014 Dec 24;15:208. doi: 10.1186/s12875-014-0208-3. PMID 25539989